CLINICAL TRIAL: NCT00964340
Title: A Randomized, Placebo-Controlled, Double-Blind, Clinical Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral SRT2104 Capsules Administered to Healthy Elderly Subjects for 28 Days
Brief Title: A Clinical Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral SRT2104 Capsules Administered to Healthy Elderly Subjects for 28 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 113312
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Atrophy, Muscular
MeSH Terms: conditions — Muscular Atrophy | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): The Placebo treatment group will be administered eight placebo capsules per day. Placebo will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every day, approximately 15 minutes following the consumption of a standardized meal, and subjects must wait at least 1-2hrs after dosing before consuming additional calories. Water is permitted ad libitum.
  Interventions: Drug: Placebo
- 0.5g SRT2104 (Active Comparator): The 0.5g SRT2104 treatment group will be administered 2 SRT2104 capsules with 6 matching placebo capsules, for a total of 8 capsules per day. 0.5g SRT2104 will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every day, approximately 15 minutes following the consumption of a standardized meal, and subjects must wait at least 1-2hrs after dosing before consuming additional calories. Water is permitted ad libitum.
  Interventions: Drug: Placebo; Drug: SRT2104
- 2.0g SRT2104 (Active Comparator): The 2.0g SRT2104 treatment group will be administered 8 SRT2104 capsules per day. 2.0g SRT2104 will be administered orally once daily for twenty-eight consecutive days. Dosing will take place at approximately the same time every day, approximately 15 minutes following the consumption of a standardized meal, and subjects must wait at least 1-2hrs after dosing before consuming additional calories. Water is permitted ad libitum.
  Interventions: Drug: SRT2104

INTERVENTIONS:
Drug: Placebo — For the placebo product, the SRT2104 drug substance will be replaced by microcrystalline cellulose (Avicel® PH 105) to match the SRT2104 investigational product. The ratio of active to placebo capsules will vary according to the subject's dosing level.
  Arms: 0.5g SRT2104; Placebo
Drug: SRT2104 — SRT2104 drug substance is a new chemical entity which is supplied as a fine, yellowish/amber powder. The SRT2104 investigational product is prepared by packing 250 mg of the SRT2104 powder into a size 00 opaque capsule, which is then stored in dosing bottles.
  Arms: 0.5g SRT2104; 2.0g SRT2104

SUMMARY:
The primary objective is to determine the pharmacokinetics, safety and tolerability of SRT2104 in healthy elderly subjects following single and 28 days dosing.

The secondary objectives of the study are:

1. To contrast changes in leg muscle function following repeat doses of SRT2104 or placebo:

   Endurance exercise tolerance 31P MRS measures of mitochondrial oxidative capacity in the gastrocnemius muscle
2. To test for a change in the ratio of visceral to subcutaneous body fat following repeat doses of SRT2104 relative to placebo using MRI
3. To estimate any changes in insulin sensitivity (using mOGTT) following repeat doses of SRT2104 or placebo
4. To test for dose-related effects on the exploratory pharmacodynamic measures above

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel group, placebo-controlled study of healthy 60-80 year old community-dwelling male and female subjects. The study consists of 8 outpatient clinic visits, 2 inpatient clinic visits and 8 telephone contacts (including the pre-screening call to determine a subject's interest in participation).

Subjects will undergo a preliminary telephone pre-screening assessment to determine their interest in participating in the study. Once interest has been confirmed, subjects will sign an informed consent and undergo screening procedures. Subjects meeting the inclusion and exclusion criteria will be enrolled in the study and randomized to receive either 0.5 g/day of SRT2104, 2.0 g/day of SRT2104 or placebo once daily for up to 28 consecutive days. After the completion of the screening assessments and confirmation of eligibility, subjects will return to the site on Day -9 and will undergo a practice endurance testing session. In addition, on Day -9 subjects will be given a pedometer which they will be asked to wear while awake for 7 consecutive days from Day -8 and 7 consecutive days from Day 20 to estimate daily physical mobility levels in the home environment. Subjects will return to the site on Days -1 and 27 for safety assessments, MRI/MRS assessments and exercise endurance tests.

On Days 1 and 28 subjects will be admitted overnight as inpatients. PK samples will be collected through 24 hours post-dose on Days 2 and 29.

During the dosing period safety visits will be performed on approximately Days 7, 14, and 21. Additional telephone safety assessments will be made approximately on Days 3, 5, 10, 17, 20 and 24.

The End of Dosing Follow-up visit will be performed approximately 35 days following the first dose of SRT2104 or placebo. An additional follow up safety telephone call will be made to each subject 30 days following their final dose of SRT2104 and/or placebo. The end of the study is defined as the last subject's last assessment (i.e. Day 58, the date of the last subject communication).

Subjects will be instructed to self administer test material at home on study days 3-27. All study visits are outpatient visits except for Day 1 and Day 28. Subjects will stay overnight at the site the evening of Day 1 and Day 28. On Day 2 and Day 29 subjects will be discharged home following the completion of study assessments and when considered clinically appropriate by the study physician.

ELIGIBILITY:
Inclusion Criteria:

* Independently ambulatory, healthy male and female subjects within the age range of 60 to 80 years (inclusive) at the time of screening
* All female subjects must be of non-childbearing potential. For the purposes of this study, women need to be amenorrheic for at least 12 consecutive months, at least 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy) or post tubal ligation. Menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 40 - 138 mIU/ml and oestradiol <20 pg/ml at entry. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH and/or oestradiol levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at the discretion of the Principal Investigator with agreement of the independent Medical Monitor
* All male subjects must agree with their partners to use double-barrier birth control or abstinence while participating in the study and for 12 weeks following the last dose of study drug
* Willingness to provide written informed consent to participate in the study
* Body Mass Index (BMI) 18-30 kg/m^2 (inclusive)
* No prior history of HIV 1 or 2
* No prior history of disease markers for hepatitis B & C virus
* Absence of significant disease or clinically significant abnormal laboratory values on the laboratory evaluations, medical history or physical examination during screening; normal end organ function at the discretion of the Principal Investigator
* Have a normal 12-lead ECG or one with changes considered to be clinically insignificant on medical review. QTcF must be <430msec for males and <450msec for females
* Resting supine BP <160/90 mmHg.
* Comprehension of the nature and purpose of the study and compliance with the requirement of the entire protocol
* Able to communicate in person and by telephone in a manner that allows all protocol procedures to be carried out safety and reliably in the opinion of the investigative site staff
* Able to take 8 capsules of study medication

Exclusion Criteria:

* Limitation to free passive or active movement of leg or foot by pain, prior injury, or developmental abnormality
* Any major illness in the past three months or any ongoing chronic medical illness which in the opinion of the PI or Medical Monitor could risk subject safety or interpretation of the results
* Ongoing or chronic history of renal or liver impairment, defined as serum creatinine clearance level less than 80ml/min as determined by Cockcroft-Gault formula (adjusted for ideal body weight), and greater than two times the upper limit of normal for liver enzymes, respectively
* Subjects with a CPK> upper limit of normal. CPK values that are marginally above the upper limit of normal may be retested at the discretion of the Principal Investigator in conjunction with the Sponsor's approval
* History, within 3 years, of drug abuse (including but not limited to anxiolytics or pain medication)
* History of alcoholism (more than two years), drinkers of more than three units per day (one unit of alcohol is equivalent to one small glass of wine, half pint of beer or one measure of spirit)
* Participation in any clinical trial with an investigative medicinal product within the past three months prior to the first dose in the current study
* Exposure to more than three new chemical entities within 12 months prior to the first dose in the current study
* History of difficulty in donating blood or accessibility of veins in left or right arm
* Donation of blood (one unit or 350 ml) within three months prior to receiving the first dose of test material
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation
* Ongoing, or history of endocrine, inflammatory, cardiovascular (in particular cardiac hypertrophy or cardiac dysrrhythmia, cardiac failure or history of prolonged QT interval), gastro-intestinal (except for appendectomy), neurological, psychiatric or metabolic disease which in the opinion of the Investigator or Medical Monitor could risk subject safety or interpretation of the results
* Active neoplastic disease or history of neoplastic disease (except for basal cell carcinoma of the skin)
* Contraindications to MRI including, but not limited to: intracranial aneurism clips (except Sugita), history of metal lathe work or possibility of intra-orbital metal fragments, pacemakers and non-MR compatible heart valves or other non-MR compatible implants, history of claustrophobia or subject feels unable to lie still on their back for a period of 1 hour in the MRI scanner
* Subjects receiving steroids, estrogens insulin or creatine will be excluded. Other concomitant medications and herbal products administered in a stable dose for at least 3 months may be permitted at the discretion of the Principal Investigator
* Subjects who spend less than 1 hour per week walking outside the home and subjects who participate in light sports and exercise for more than 6 hours per week
* A positive pre-study drug/alcohol screen
* Ongoing, or history of Type 1 or Type 2 diabetes mellitus or mOGTT results at screening that in the opinion of the PI indicates diabetes or pre-diabetes

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2010-04-27 (Actual); Study Completion 2010-04-27 (Actual)

PRIMARY OUTCOMES:
Determine the pharmacokinetics of SRT2104 in healthy elderly subjects following single and 28 days dosing. | PK samples will be collected on Days 1 and 28 at pre-dose and at 15 min, 30 min, and 1, 2, 3, 4, 8, 12 hrs post-dose. PK samples will also be collected 24 hrs post-dose on Days 2 and 29.
Safety and tolerability of SRT2104 in healthy elderly subjects following single and 28 days dosing. | Safety will be monitored by AEs, VS, physical exam, labs and ECGs during the study.

SECONDARY OUTCOMES:
Contrast changes in leg muscle function following repeat doses of SRT2104. | On Day -1 and Day 27, 31P MRS will measure mitochondrial oxidative capacity in the gastrocnemius muscle of the dominant leg; exercise in the MR scanner and a staged bicycle exercise test will record the exercise endurance tolerance.
Test for a change in the ratio of visceral to subcutaneous body fat by MRI following repeat doses of SRT2104 or placebo. | On Day -1 and Day 27 MRI and MRS assessments will be performed to measure compartmental fat distribution.
Measure changes in insulin sensitivity (using mOGTT) and dose-related effects on pharmacodynamics following repeat doses of SRT2104 or placebo. | OGTT is measured to assess PD effects of SRT2104 at screening and on Day 29 prior to the administration of 75g of oral glucose, and at 10min, 20min, 30min, 1hr, 1.5hr, 2hr, and 3 hr following glucose administration.
Test for an increase in overall endurance and activity following repeat doses of SRT2104. | Pedometer will be worn by subjects while awake for 7 consecutive days from Day -8 until Day -1 and on Day 20 until Day 27.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Libri V, Brown AP, Gambarota G, Haddad J, Shields GS, Dawes H, Pinato DJ, Hoffman E, Elliot PJ, Vlasuk GP, Jacobson E, Wilkins MR, Matthews PM. A pilot randomized, placebo controlled, double blind phase I trial of the novel SIRT1 activator SRT2104 in elderly volunteers. PLoS One. 2012;7(12):e51395. doi: 10.1371/journal.pone.0051395. Epub 2012 Dec 20. PMID 23284689
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113312 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113312?search=study&study_ids=113312#rs
- Available data/document: Informed Consent Form: 113312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113312 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register